CLINICAL TRIAL: NCT06270602
Title: A Retrospective-prospective, Observational, Multicentric Study to Record Data From the ROC Platform and Monitor the ROC Performance
Brief Title: The ONCOCAMP Study
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: ONCOCAMP; 6/23 oss (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2024-01-29; First posted 2024-02-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Oncology
Keywords: Oncological Network; Multidisciplinary Oncology Groups
MeSH Terms: conditions — Neoplasms | interventions — Data Collection; Retrospective Studies; Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (Retrospective):: All consecutive patients entered in the ROC platform from the start of platform activation (November 2018) until the date in which the study is approved by the local ethical committee (Investigator is allowed to enroll patients) will be enrolled. The retrospective cohort will be made by more than 40000 patients already included in the platform and entered a GOM path
  Interventions: Other: Data collection (retrospective)
- Cohort B (Prospective):: All consecutive patients who enter in the ROC platform as for clinical practice from the date in which the study is approved by the local ethical committee (Investigator is allowed to enroll patients).
  Interventions: Other: Data collection (prospective)

INTERVENTIONS:
Other: Data collection (retrospective) — Collection of patient data entered in the ROC platform from the beginning activation of the platform (November 2018) until the date on which the study is approved by the local ethics committee
  Groups: Cohort A (Retrospective):
Other: Data collection (prospective) — Collection of patient data entered in the ROC platform from the date in which the study is approved by the local ethical committee
  Groups: Cohort B (Prospective):

SUMMARY:
The present study is a retrospective-prospective observational and multicentric study aiming to collect data relating to all patients included in the ROC platform. All ROC centers will be involved in the present study.

DETAILED DESCRIPTION:
The ROC platform therefore represents a multicenter database and a growing source of data and information regarding cancer patients in the Campania region. The need for multicenter databases is supported by the results obtained with both retrospective and prospective studies. Many retrospective studies have led to changes in some of the available guidelines. Important advantages of this study include representativeness of the analyzed cohort to all patients with a specific cancer and a large sample size that provides sufficient statistical power to detect differences across different patient groups. The data extracted from the ROC have the potential to produce knowledge, to guide decision-making, and to manage more effectively the challenges of fighting cancer in our region. The Campania region counts more than 6 million people, and it is characterized by a worst oncological outcome compared to the average data of other Italian region: the ROC platform has the potential to analyze the effect of a public intervention in the field of oncology care. Therefore, the primary aim of this study is to create a retrospective-prospective registry of all cancer patients entering the ROC platform and in a GOM path describing the primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* registration in the ROC platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All consecutive patients entered in the ROC platform from the start of platform activation (November 2018) until the date in which the study is approved by the local ethical committee (The retrospective cohort will be made by more than 40000 patients already included in the platform and entered a GOM path.
  2. All consecutive patients who enter in the ROC platform as for clinical practice from the date in which the study is approved by the local ethical committee (Investigator is allowed to enroll patients).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence for each tumor of the patients included in the ROC platform | Every year up to 5 years
  Incidence for each tumor of the patients included in the ROC platform
Evaluation of the time interval between GOM activities | Every 6 months up to 3 years
  Time interval between reporting and taking charge by the GOM, the date diagnosis and the GOM meeting date, the first GOM meeting and the final therapeutic decision, the therapy decision and the therapeutic act, and the request for home assistance and the actual taking in charge by the ASL
Evaluation of the time interval between GOM activities | Every 6 months up to 3 years
  Time interval between the request for home assistance and the actual taking in charge by the ASL
Evaluation of the time interval between GOM activities | Every 6 months up to 3 years
  Time interval between the therapy decision and the therapeutic act
Evaluation of the time interval between GOM activities | Every 6 months up to 3 years
  Time interval between the first GOM meeting and the final therapeutic decision
Evaluation of the time interval between GOM activities | Every 6 months up to 3 years
  Time interval betweenthe date diagnosis and the GOM meeting date
Frequency of use of the services of the ROC platform | Every 2 months up to 5 years
  Frequency of use of the services of the ROC platform
Descriptive analysis of each subgroup of patients (subdivision by tumor type) | Every 6 months up to 5 years
  Descriptive analysis of each subgroup of patients (subdivision by tumor type)
Spatial analysis for each patient | Every year up to 5 years
  Spatial analysis for each patient
Frequency of adherence to guidelines of the Diagnostic Therapeutic Assistance Paths (PDTA) | Every 6 months up to 5 years
  Frequency of adherence to guidelines of the Diagnostic Therapeutic Assistance Paths (PDTA)
Percentage of patient included in clinical trial | Every 2 months up to 5 years
  Percentage of patient included in clinical trial
Assessment of costs arising due to inefficiencies (repetition and inappropriateness of diagnostic tests; passive health mobility rate | Every 6 months up to 5 years
  Assessment of costs arising due to inefficiencies (repetition and inappropriateness of diagnostic tests; passive health mobility rate
Prevalence for each tumor of the patients included in the ROC platform | Every year up to 5 years
  Prevalence for each tumor of the patients included in the ROC platform

SECONDARY OUTCOMES:
Description of pharmacological strategies | Every year up to 5 years
  Evaluation of pharmacological strategies
Description of diagnostic activities | Every year up to 5 years
  Evaluation of diagnostic activities
Description of surgical strategies | Every year up to 5 years
  Evaluation of surgical strategies
Appropriateness of diagnostic tests (taking as reference the guidelines reported in each PDTA) | Every 6 months up to 5 years
  Appropriateness of diagnostic tests (taking as reference the guidelines reported in each PDTA)
Description of each surgical approach | Every year up to 5 years
  Description of each surgical approach
Description of the different surgical techniques among the centers | Every year up to 5 years
  Description of the different surgical techniques among the centers
Patients' quality of life | Every year up to 5 years
  Patients' quality of life using questionnaires
Patients' reported outcome | Every year up to 5 years
  Patients' reported outcome using questionnaires
Patients' satisfaction and evaluation of the diagnostic / therapeutic path | Every year up to 5 years
  Patients' satisfaction and evaluation of the diagnostic / therapeutic path using questionnaires
Correlation analysis among risk factors and diagnostic / therapeutic delay or poor prognosis | Every year up to 5 years
  Correlation analysis among risk factors and diagnostic / therapeutic delay or poor prognosis
Dependence analysis between the conditions of social deprivation of ROC patients and the time to the first GOM visit | Every year up to 5 years
  Dependence analysis between the conditions of social deprivation of ROC patients and the time to the first GOM visit
Dependence analysis among costs, socio-demographic characteristics and some variables related to the diagnostic / therapeutic path | Every year up to 5 years
  Dependence analysis among costs, socio-demographic characteristics and some variables related to the diagnostic / therapeutic path
Survival analysis for each tumor | Every 2 years up to 6 years
  Survival analysis for each tumor
Life status assessment for each patient | Every year up to 5 years
  Life status assessment for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (17):
- Italy (17):
  - A.O. Moscati, Avellino, Avellino
  - Asl Avellino, Avellino, Avellino
  - A.O. Rummo, Benevento, Benevento
  - Asl Benevento, Benevento, Benevento
  - Asl Caserta, Caserta, Caserta
  - A.O. S.Anna S. Sebastiano, Caserta, Caserta
  - Asl Napoli 2 Nord, Casavatore, Napoli
  - Asl Napoli 3 Sud, Ercolano, Napoli
  - A.O. Cardarelli, Napoli, Napoli
  - A.O. Dei Colli, Napoli, Napoli
  - Federico II, Napoli, Napoli
  - I.N.T. Pascale, Napoli, Napoli
  - A.O.U. Luigi Vanvitelli, Napoli, Napoli
  - Asl Napoli 1 Centro, Napoli, Napoli
  - Ospedale del Mare, Napoli, Napoli
  - Asl Salerno, Salerno, Salerno
  - A.O.U. Ruggi, Salerno, Salerno

REFERENCES:
- [Derived] Porciello G, Di Lauro T, Luongo A, Coluccia S, Prete M, Abbadessa L, Coppola E, Di Martino A, Mozzillo AL, Racca E, Piccirillo A, Di Giacomo V, Fontana M, D'Amico M, Palumbo E, Vitale S, D'Errico D, Turra V, Parascandolo I, Stallone T, Augustin LSA, Crispo A, Celentano E, Pignata S. Optimizing Nutritional Care with Machine Learning: Identifying Sarcopenia Risk Through Body Composition Parameters in Cancer Patients-Insights from the NUTritional and Sarcopenia RIsk SCREENing Project (NUTRISCREEN). Nutrients. 2025 Apr 18;17(8):1376. doi: 10.3390/nu17081376. PMID 40284239